CLINICAL TRIAL: NCT03123796
Title: Effects of Proton Pump Inhibitors on Kidney Transplant Recipients
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Yasar Caliskan, Associate Professor of Medicine, Istanbul University
Other Study IDs: 332
Record Dates: First submitted 2017-04-19; First posted 2017-04-21 (Actual); Last update posted 2017-12-27 (Actual); Status verified 2017-12

CONDITIONS: Transplant Dysfunction; Magnesium Disorder
Keywords: chronic rejection; transplant outcome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Only PPI: Kidney transplant recipients who used only proton pump inhibitors and did not use histamine H2 receptor antagonists.
- Only H2RA: Kidney transplant recipients who used only histamine H2 receptor antagonists and did not use proton pump inhibitors.
- PPI and H2RA: Kidney transplant recipients who used both proton pump inhibitors and histamine H2 receptor antagonists.
- No Acid Suppressive Treatment: Kidney transplant recipients who used neither proton pump inhibitors nor histamine H2 receptor antagonists.

SUMMARY:
Use of proton pump inhibitors (PPIs) is quite common among renal transplant recipients and reduced kidney functions and hypomagnesemia with the use of PPIs have been reported. In this study, investigation of the effects of PPI use on the outcome of kidney transplant recipients is aimed.

DETAILED DESCRIPTION:
Use of proton pump inhibitors (PPIs) is frequent among renal transplant recipients due to the common use of glucocorticoids in immunosuppresive regimens after transplantation. Reduced kidney functions and hypomagnesemia with the use of PPIs have been reported in various patient populations. However, few studies examined the effects of PPIs on kidney transplant recipients. Therefore, the aim of this study is to investigate the effects of PPI and/or histamine H2 receptor antagonist use on serum magnesium levels, allograft functions and survival in kidney transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant recipients who used only proton pump inhibitors and did not use histamine H2 receptor antagonists (Only PPI).
* Kidney transplant recipients who used histamine H2 receptor antagonists and did not use proton pump inhibitors (Only H2RA).
* Kidney transplant recipients who used both proton pump inhibitors and histamine H2 receptor antagonists (PPI and H2RA).
* Kidney transplant recipients who used neither proton pump inhibitors nor histamine H2 receptor antagonists (No Acid Suppressive Treatment).

Exclusion Criteria:

* Patients who are unwilling or unable to consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kidney transplant recipients.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Graft survival | 5-10 years

SECONDARY OUTCOMES:
Graft rejection | 5-10 years

OTHER OUTCOMES:
Serum magnesium levels | 5-10 years

CONTACTS AND LOCATIONS:
Overall Officials: Yasar Caliskan, MD, Principal Investigator — Division of Nephrology, Department of Internal Medicine, Istanbul Faculty of Medicine
Locations (1):
- Division of Nephrology, Department of Internal Medicine, Istanbul Faculty of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lazarus B, Chen Y, Wilson FP, Sang Y, Chang AR, Coresh J, Grams ME. Proton Pump Inhibitor Use and the Risk of Chronic Kidney Disease. JAMA Intern Med. 2016 Feb;176(2):238-46. doi: 10.1001/jamainternmed.2015.7193. PMID 26752337
- [Background] van Boekel GA, Kerkhofs CH, van de Logt F, Hilbrands LB. Proton pump inhibitors do not increase the risk of acute rejection. Neth J Med. 2014 Feb;72(2):86-90. PMID 24659591